CLINICAL TRIAL: NCT05951088
Title: Long-term Evaluation of a Mobile Application for Follow-up of Cardiac Patients
Brief Title: Long-term Evaluation of a Mobile Application for Follow-up of Cardiac Patients (Cardio2U Study)
Acronym: Cardio2U
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Other Study IDs: BUN B3002023000007
Record Dates: First submitted 2023-06-15; First posted 2023-07-18 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-03

CONDITIONS: Follow-up; Education; Mobile Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- atrial fibrillation patients: AF patients hospitalised at the cardiology department or coming for an outpatient visit
  Interventions: Procedure: Cardio2U follow-up
- heart failure patients: HF patients hospitalised at the cardiology department or coming for an outpatient visit
  Interventions: Procedure: Cardio2U follow-up

INTERVENTIONS:
Procedure: Cardio2U follow-up — During the follow-up period, participants will have access to the application and will be able to explore the different modules. At fixed time points, the application will allow them to fill in questionnaires about the application's usability and patient satisfaction. App user data will track how long and how often patients visit the application and which aspects are mostly used. In addition, at different time points during the study, patients will be asked to complete clinical questionnaires regarding e.g. patients' knowledge and self-care abilities. The results of these questionnaires can be used in a more clinical way as they will be accessible to doctors and nurses in the healthcare provider dashboard and can support targeted patient follow-up and guidance

SUMMARY:
This trial has to aim to evaluate an innovative, in-house developed mobile application supporting patients in their home environment by actively involving them in different aspects of their condition and treatment. The usability, long-term adherence and patient satisfaction will be studied in patients with atrial fibrillation (AF) and/or heart failure (HF).

DETAILED DESCRIPTION:
Atrial fibrillation (AF) and heart failure (HF) are global cardiovascular disease epidemics associated with significant morbidity and mortality. Their prevalence is already high and will continue to increase in the coming decades. A structured and efficient care system encompassing various aspects is needed to manage AF and HF morbidity and mortality. Technological developments and the increased use of smart devices, including in medical care, create opportunities to implement mobile applications to provide continuous, high-quality follow-up to patients. Our in-house developed application, recently improved and expended, provides a reliable source of educational material on AF and HF, with the ability to save health appointments, enter measurements (such as heart rate, blood pressure, weight) and keep a medication list (including notifications when medication should be taken). In addition, the application includes questionnaires to assess, for example, patients' knowledge, selfcare, quality of life, physical activity and symptoms. The application allows personalisation per patient depending on the clinical setting and indication. The innovative application will be evaluated in terms of usability, long-term adherence and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years,
2. Patients in whom AF or atrial flutter is diagnosed with an electrocardiogram (12-lead, Holter monitor,…) and/or patients in whom HF is diagnosed in their medical records,
3. Patients who are capable of signing the informed consent.

Exclusion Criteria:

1. Not able to speak and read Dutch,
2. Cognitive impaired (e.g. severe dementia),
3. No smartphone or tablet available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AF and/or HF hospitalised at the cardiology department or coming for an outpatient visit, will be asked to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Usability of the application | Change of usabilitiy of the application from baseline to12 months
  Usability will be evaluated during the follow-up period using a specific 'Usability Questionnaire'.
Patient satisfaction with the application-driven follow-up | Change from baseline patient satisfaction with the application to 3- and 12 months
  Patient satisfaction will be evaluated during the follow-up period using a specific 'Satisfaction Questionnaire'.
Long-term adherence | From date of randomization until end of study, assessed up to 36 months
  Long-term adherence will be measured using the app user data

SECONDARY OUTCOMES:
Disease specific Knowledge | Change from baseline to 1, 3, 6, and 12 months
  Patients knowledge about AF and its treatment will be assessed during their follow-up using disease specific knowledge questionnaires
Disease specific self-care management | Change from baseline to 3 and 12 months
  Patients self-care possibilities will be assessed during their follow-up using a specific self-care questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Hein Heidbuchel, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium